CLINICAL TRIAL: NCT07182500
Title: The Effect of Bifidobacterium Probiotics on Gut Microbiota Changes in Healthy Adults During Short-term Travel Along the Silk Road
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Collaborators: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Min-Tze LIONG, Prof., Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SJUPN-2025-013-HY1-KS2
Record Dates: First submitted 2025-09-08; First posted 2025-09-19 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Healthy Adult Volunteer
Keywords: probiotc; travel; Silk Road
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Daily 6-drops of non-GMO corn starch in medium-chain triglyceride oil
  Interventions: Other: Placebo
- Probiotic (Experimental): Daily 6-drops of Bifidobacterium longum subsp. infantis M-63, B. breve M-16V, and B. longum BB536 in non-GMO corn starch as excipient, in medium-chain triglyceride oil (1.5 × 109 CFU/day)
  Interventions: Other: Probiotic

INTERVENTIONS:
Other: Probiotic — Daily 6-drops of Bifidobacterium longum subsp. infantis M-63, B. breve M-16V, and B. longum BB536 in non-GMO corn starch as excipient, in medium-chain triglyceride oil (1.5 × 109 CFU/day)
  Arms: Probiotic
Other: Placebo — Daily 6-drops of non-GMO corn starch in medium-chain triglyceride oil
  Arms: Placebo

SUMMARY:
Journeying along the historic Silk Road exposes travelers to dramatic dietary shifts, unfamiliar microbial environments, and the physical stresses of long-distance travel-all known to disrupt gut health and cause gastrointestinal complaints, including traveler's diarrhea and sleep disturbances. Such disruptions may also elevate the risk of acquiring antibiotic-resistant organisms.

This randomized, double-blind, placebo-controlled trial evaluated whether probiotic supplementation can help maintain gut microbial balance and support traveler well-being during trips to Silk Road regions. In addition to monitoring changes in gut microbiota composition, the study assessed gastrointestinal symptoms, sleep quality, anxiety levels, overall well-being, gut immune markers, functional profiles of the microbiome, and the presence of antibiotic resistance genes.

DETAILED DESCRIPTION:
Journeys along the Silk Road-with their unique dietary shifts, unfamiliar water and food sources, novel microbial exposures, altered sleep patterns, and psychological adjustments-can significantly disrupt gut microbiota and impact overall health. Prior research has shown that even short-term travel can lead to substantial fluctuations in gut microbial composition, often accompanied by gastrointestinal symptoms and reduced well-being, underscoring the need for effective strategies to support gut homeostasis during such journeys.

Gastrointestinal distress, including traveler's diarrhea and non-diarrheal symptoms such as abdominal pain and irregular bowel movements, remains a common challenge. These issues can considerably diminish the travel experience. Furthermore, travel has been linked to an elevated risk of acquiring antimicrobial resistance genes, with the gut serving as a potential site for the exchange and amplification of resistant organisms.

Sleep disruptions-stemming from changes in routine and environment-also play an important role in traveler well-being. The gut-brain axis provides a mechanism through which sleep quality may influence gastrointestinal vulnerability, highlighting the interconnected nature of these systems.

Probiotics represent a promising intervention to support travelers. These beneficial microorganisms may enhance gut barrier function, modulate immune activity, inhibit pathogens, and produce metabolites that contribute to both gut and systemic health. Although some studies suggest probiotics can alleviate gastrointestinal symptoms and reduce the risk of diarrhea, robust evidence specific to the Silk Road travel context remains limited.

In this randomized, double-blind, placebo-controlled trial, effects of daily probiotic supplementation on gut microbiota stability, gastrointestinal symptoms, sleep quality, anxiety, and overall well-being in adults traveling the Silk Road will be evaluated. Immune markers, microbial functional pathways, and antibiotic resistance gene profiles will be identified to better understand the potential mechanisms of action. The investigators hypothesized that probiotic intake would help maintain microbial balance, reduce travel-related symptoms, and support physical and emotional well-being throughout the journey.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy adults
* Scheduled to undertake a short-term round trip (less than 7 days) to abroad
* Able to complete study procedures
* Willing to take intervention products

Exclusion Criteria:

* Use of antibiotics, probiotics, hormones, immunosuppressants, biologics or JAK inhibitors within four weeks prior to study
* Chronic or severe systemic diseases (including cardiovascular, hepatic, renal, malignant or psychiatric disorders)
* Uncontrolled parasitic infections
* Long-term use of corticosteroids, growth hormone, vitamin B12, lysine or inositol
* Major surgery within one month
* Allergy to probiotic components
* Other conditions deemed inappropriate by investigators

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-10-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Microbiota profiles of fecal samples in generally healthy adults upon administration of probiotic as assessed via metagenomics sequencing | 7 days
  Differences in microbiota abundance in fecal sample of generally healthy adults upon administration of probiotic as compared to placebo

SECONDARY OUTCOMES:
Respiratory symptoms duration and frequency in generally healthy adults upon administration of probiotic as assessed using questionnaire | 7 days
  Changes in duration and frequency of respiratory illnesses symptoms from generally healthy adults on probiotic or placebo after 7-days, via the use of standard clinical assessment questionnaire, scale 0-3 where higher scores indicate more severe symptoms
Gastrointestinal symptoms in generally healthy adults upon administration of probiotic as assessed using questionnaire | 7 days
  Differences in duration and frequency of gastrointestinal symptoms upon administration of probiotic compared to placebo via the use of standard clinical assessment questionnaire, scale 0-3 where higher scores indicate more severe symptoms
Allergy symptoms in generally healthy adults upon administration of probiotic as assessed using questionnaire | 7 days
  Differences in duration and frequency of allergy symptoms upon administration of probiotic compared to placebo via the use of standard clinical assessment questionnaire, scale 0-3 where higher scores indicate more severe symptoms
Gastrointestinal metabolites in generally healthy adults upon administration of probiotic as assessed using LC-MS | 7 days
  Differences in concentrations of gastrointestinal metabolites upon administration of probiotic compared to placebo
Anxiety in generally healthy adults upon administration of probiotic as assessed using questionnaire | 7 days
  Differences in anxiety via the GAD-7 questionnaire （scale 0-3 where higher scores indicate more severe outcomes), upon administration of probiotic compared to placebo
Sleep quality in generally healthy adults upon administration of probiotic as assessed using questionnaire | 7 days
  Differences in sleep quality via the PSQI questionnaire （scale 0-3 where higher scores indicate more severe outcomes) upon administration of probiotic compared to placebo
Well-being in generally healthy adults upon administration of probiotic as assessed using questionnaire | 7 days
  Differences in well-being via the WHO-5 questionnaire (scale 0-5 where higher scores indicate better outcomes）upon administration of probiotic compared to placebo

CONTACTS AND LOCATIONS:
Overall Officials: Meiqin Cai, MD., Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (2):
- Shanghai Jiao Tong University School of Medicine, Huangpu, Shanghai Municipality, China
- Universiti Sains Malaysia, George Town, Pulau Pinang, Malaysia

IPD SHARING:
Plan to Share IPD: No